CLINICAL TRIAL: NCT02322281
Title: TIGER-3: A Phase 3, Open-label, Multicenter, Randomized Study of Oral Rociletinib (CO-1686) Monotherapy Versus Single-agent Cytotoxic Chemotherapy in Patients With Mutant EGFR Non-small Cell Lung Cancer (NSCLC) After Failure of at Least 1 Previous EGFR-directed Tyrosine Kinase Inhibitor (TKI) and Platinum-doublet Chemotherapy
Brief Title: TIGER-3: Open Label, Multicenter Study of Rociletinib (CO-1686) Mono Therapy Versus Single-agent Cytotoxic Chemotherapy in Patients With Mutant EGFR NSCLC Who Have Failed at Least One Previous EGFR-Directed TKI and Platinum-doublet Chemotherapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor discontinued development of CO-1686 for NSCLC
Sponsor: Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO-1686-020 (TIGER-3)
Record Dates: First submitted 2014-12-17; First posted 2014-12-23 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: cancer; metastatic; locally advanced; lung; non-small cell lung cancer; NSCLC; epidermal growth factor receptor; EGFR; T790M; CO-1686; unresectable; recurrent; EGFR-directed therapy; irreversible EGFR inhibitor; TIGER; Rociletinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Neoplasm Metastasis; Recurrence | interventions — rociletinib; Pemetrexed; Gemcitabine; Paclitaxel; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rociletinib Monotherapy (500 mg BID) (Experimental): Daily oral rociletinib at 500 mg BID with 8 oz (240 mL) of water and with a meal or within 30 minutes after a meal. Treatment with rociletinib is continuous and each cycle will comprise of 21 days.
  Interventions: Drug: Rociletinib
- Rociletinib Monotherapy (625 mg BID) (Experimental): Daily oral rociletinib at 625 mg BID with 8 oz (240 mL) of water and with a meal or within 30 minutes after a meal. Treatment with rociletinib is continuous and each cycle will comprise of 21 days.
  Interventions: Drug: Rociletinib
- Pemetrexed or gemcitabine or paclitaxel or docetaxel (Active Comparator): Pemetrexed
  500 mg/m2 pemetrexed given intravenously on Day 1 of each 21-day cycle.
  Gemcitabine
  1250 mg/m2 gemcitabine given intravenously on Day 1 and 8 of each 21-day cycle.
  Docetaxel
  75 mg/m2 docetaxel (60 mg/m2 for patients residing in East-Asian territories) given intravenously on Day 1 of each 21-day cycle.
  or 35 mg/m2 docetaxel given intravenously on a weekly basis as part of a continuous 21-day cycle; i.e. dosing will be on Days 1, 8, and 15 of each 21-day cycle.
  Paclitaxel
  80 mg/m2 paclitaxel given intravenously on a weekly basis as part of a continuous 21-day cycle; i.e. dosing will be on Days 1, 8, and 15 of each 21-day cycle.
  Interventions: Drug: Pemetrexed or gemcitabine or paclitaxel or docetaxel

INTERVENTIONS:
Drug: Rociletinib
  Other Names: CO-1686
  Arms: Rociletinib Monotherapy (500 mg BID); Rociletinib Monotherapy (625 mg BID)
Drug: Pemetrexed or gemcitabine or paclitaxel or docetaxel
  Arms: Pemetrexed or gemcitabine or paclitaxel or docetaxel

SUMMARY:
The purpose of this study is to compare the anti-tumor efficacy of oral single-agent rociletinib, as measured by investigator assessment of the PFS, with that of single-agent cytotoxic chemotherapy in patients with EGFR-mutated, advanced/metastatic NSCLC after failure of at least 1 previous EGFR-directed TKI and at least 1 line of platinum-containing doublet chemotherapy.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, open-label, multicenter study evaluating the safety and efficacy of oral rociletinib at 500 mg BID and 625 mg BID compared with that of single-agent cytotoxic chemotherapy, in patients with previously treated mutant EGFR NSCLC. Eligible patients are those with mutant EGFR NSCLC previously treated with at least 1 EGFR inhibitor and at least 1 line of platinum-containing chemotherapy doublet for advanced/metastatic NSCLC.

After providing informed consent to participate and screening to confirm eligibility, patients will be randomized 1:1:1 to receive either oral rociletinib 500 mg BID, oral rociletinib 625 mg BID, or single-agent cytotoxic chemotherapy (investigator choice of pemetrexed, gemcitabine, docetaxel, or paclitaxel; choice of chemotherapy agent must be specified before randomization).

ELIGIBILITY:
Inclusion Criteria:

All patients must meet all of the following inclusion criteria:

1. Histologically or cytologically confirmed metastatic or unresectable locally advanced NSCLC with radiological progression on the most recent therapy received
2. Documented evidence of a tumor with 1 or more EGFR activating mutations excluding exon 20 insertion
3. Disease progression confirmed by radiological assessment while receiving treatment with single agent EGFR-TKI (e.g., erlotinib, gefitinib, afatinib, or dacomitinib) or EGFR-TKI in combination with other targeted therapy (e.g. bevacizumab, immunotherapy)
4. Multiple lines of prior treatment are permitted and there is no specified order of treatment, but in the course of their treatment history, patients must have received and have radiologically documented disease progression following:

   At least 1 line of prior treatment with a single-agent EGFR-TKI (e.g., erlotinib, gefitinib, afatinib, or dacomitinib)

   If EGFR-TKI is a component of the most recent treatment line, the washout period for the EGFR-TKI is a minimum of 3 days before the start of study drug treatment

   AND

   A platinum-containing doublet chemotherapy (either progressed during therapy or completed at least 4 cycles without progression with subsequent progression after a treatment-free interval or after a maintenance treatment).

   If cytotoxic chemotherapy is a component of the most recent treatment line, treatment with chemotherapy should have been completed at least 14 days prior to start of study treatment. When an EGFR-TKI is given in combination with platinum-containing doublet chemotherapy, treatment with the EGFR-TKI may continue until at least 3 days before start of treatment.
5. Have undergone a biopsy of either primary or metastatic tumor tissue within 60 days prior to start of treatment and have tissue sent to the central laboratory prior to randomization
6. Measureable disease according to RECIST Version 1.1
7. Life expectancy of at least 3 months
8. ECOG performance status of 0 to 1
9. Age ≥ 18 years (in certain territories, the minimum age requirement may be higher e.g., age ≥ 20 years in Japan and Taiwan, age ≥ 21 years in Singapore)
10. Patients should have recovered to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade ≤ 1 from any significant chemotherapy-related toxicities
11. Adequate hematological and biological function
12. Written consent on an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved ICF before any study specific evaluation

Exclusion Criteria:

Any of the following criteria will exclude patients from study participation:

1. Any other malignancy associated with a high mortality risk within the next 5 years and for which the patients may be (but not necessarily) currently receiving treatment

   Patients with a history of malignancy that has been completely treated, with no evidence of that cancer currently, are permitted to enroll in the trial provided all chemotherapy was completed > 6 months prior and/or bone marrow transplant > 2 years prior
2. Known pre-existing interstitial lung disease
3. Tumor small cell transformation by local assessment, irrespective of presence of T790M+ component
4. Patients with leptomeningeal carcinomatosis are excluded. Other central nervous system (CNS) metastases are only permitted if treated, asymptomatic, and stable (not requiring steroids for at least 2 weeks prior to randomization and the patient is neurologically stable i.e. free from new symptoms of brain metastases)
5. Patients who are currently receiving treatment with any medications that have the potential to prolong the QT interval and that treatment cannot be either discontinued or switched to a different medication (known to have no effect on QT) before starting protocol-specified treatment (see http://crediblemeds.org/ for a list of QT-prolonging medications)
6. Prior treatment with rociletinib, or other drugs that target T790M+ mutant EGFR with sparing of WT-EGFR including but not limited to osimertinib, HM61713, and TAS-121
7. Any contraindications for therapy with pemetrexed, paclitaxel, gemcitabine or docetaxel unless a contraindication with respect to one of these drugs will not affect the use of any of the others as a comparator to rociletinib
8. Any of the following cardiac abnormalities or history:

   1. Clinically significant abnormal 12-lead ECG, QT interval corrected using Fridericia's method (QTCF) > 450 msec
   2. Inability to measure QT interval on ECG
   3. Personal or family history of long QT syndrome
   4. Implantable pacemaker or implantable cardioverter defibrillator
   5. Resting bradycardia < 55 beats/min
9. Non-study related surgical procedures ≤ 7 days prior to randomization. In all cases, the patient must be sufficiently recovered and stable before treatment administration
10. Females who are pregnant or breastfeeding
11. Refusal to use adequate contraception for fertile patients (females and males) while on treatment and for 6 months after the last dose of study treatment (rociletinib and chemotherapy irrespective of single cytotoxic agent used)
12. Presence of any serious or unstable concomitant systemic disorder incompatible with the clinical study (e.g., substance abuse, uncontrolled intercurrent illness including uncontrolled diabetes, active infection, arterial thrombosis, and symptomatic pulmonary embolism)
13. Any other reason the investigator considers the patient should not participate in the study
14. Treatment with live vaccines initiated less than 4 weeks prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2015-02; Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (80):
- United States (31):
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - City of Hope Cancer Center, Duarte, California
  - Saint Joseph Heritage Healthcare, Fullerton, California
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Cancer Care Associates Medical Group, Inc., Redondo Beach, California
  - Sutter Cancer Center, Sacramento, California
  - University of California, San Francisco Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - University of California at Los Angeles, Santa Monica, California
  - Stanford University School of Medicine, Stanford, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - Sylvester Comprehensive Cancer Center (UMHC), Deerfield Beach, Florida
  - University of Florida Health Science Center, Gainesville, Florida
  - Memorial Healthcare System, Pembroke Pines, Florida
  - Northside Hospital, Atlanta, Georgia
  - North Shore University Health System, Evanston, Illinois
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Regional Cancer Care Associates, LLC, East Brunswick, New Jersey
  - Regional Cancer Care Associates, Morristown, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Providence Health and Services, Portland, Oregon
  - Oregon Health & Science University (OHSU) - Knight Cancer Institute, Portland, Oregon
  - University of Pittsburgh Cancer Institute (UPMC), Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
- Australia (3):
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
- France (9):
  - Hopital Hautepierre (CHU) de Strasbourg, Strasbourg, Alsace
  - Centre François Baclesse, Caen, Basse-Normandie
  - Centre Hospitalier Universitaire de Rennes, Hôpital Pontchaillou, Rennes, Brittany Region
  - CHRU de Lille - Hôpital Calmette, Lille, Hauts-de-France
  - CHRU de Limoges - Hôpital Dupuytren, Limoges, Limousin
  - L'Assistance Publique - Hopitaux de Marseille, Marseille, Provence-Alpes-Côte d'Azur Region
  - Centre Léon Bérard, Lyon
  - Centre Hospitalier Intercommunal Créteil, Créteil, Île-de-France Region
  - Hôpital Bichat-Claude Bernard, Paris, Île-de-France Region
- Germany (6):
  - Asklepios Fachkliniken München-Gauting, Gauting, Baden-Wurttemberg
  - Thoraxklinik Heidelberg gGmbH, Heidelberg, Baden-Wurttemberg
  - LMU - Klinikum der Universität München, München, Bavaria
  - Pius Hospital Oldenburg, Oldenburg, Niedersachen
  - Johannes-Wesling-Klinikum Minden, Minden, North Rhine-Westphalia
  - LungenClinic Großhansdorf GmbH, Großhansdorf, Schleswig-Holstein
- Italy (6):
  - A.O.U. San Luigi Gonzaga di Orbassano, Orbassano, Torino
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - IRCCS Azienda Ospedaliera Universitaria San Martino - IST, Genova
  - Ospedale Civile di Livorno, Livorno
  - Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliera di Perugia, Perugia
- Netherlands (3):
  - Academisch Ziekenhuis Maastricht, Maastricht, Limburg
  - Antoni van Leeuwenhoek Hospital, Amsterdam, North Holland
  - Universitair Medisch Centrum Groningen, Groningen
- South Korea (6):
  - Chungbuk National University Hospital, Cheongju-si, Cheungcheongbuk-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea Saint Vincent's Hospital, Suwon, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Spain (7):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de Mataró, Mataró, Barcelona
  - Institut Universitari Dexeus, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Fundacion Jimenez Diaz (Clinica de la Concepcion) (UAM -FJD), Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
- Taiwan (5):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng-Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (4):
  - University College London Hospitals, London, England
  - Guy's and Saint Thomas NHS Foundation Trust, London, England
  - Royal Marsden NHS Trust, London, England
  - The Christie NHS Foundation Trust, Manchester, England

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 149 subjects recruited from 83 sites in 10 countries and randomized (1:1) to treatment with rociletinib or single-agent cytotoxic chemotherapy (investigator's choice of pemetrexed, gemcitabine, docetaxel, or paclitaxel). Crossover to rociletinib treatment permitted for comparator chemotherapy treated subjects but only after eligibility confirmed.
Groups:
- Rociletinib 500 mg BID: Starting dose of 500mg. Taken orally twice daily (continuous 21 day treatment cycle). Treatment duration until radiographically confirmed disease progression.
- Rociletinib 625 mg BID: Starting dose of 625mg. Taken orally twice daily (continuous 21 day treatment cycle). Treatment duration until radiographically confirmed disease progression.
- Chemotherapy: Pemetrexed - 500 mg/m2 pemetrexed given intravenously on Day 1 of each 21-day cycle.
  Gemcitabine - 1250 mg/m2 gemcitabine given intravenously on Day 1 and 8 of each 21-day cycle.
  Paclitaxel - 80 mg/m2 paclitaxel given intravenously on a weekly basis as part of a continuous 21-day cycle; i.e. dosing will be on Days 1, 8, and 15 of each 21-day cycle.
  Docetaxel - 75 mg/m2 docetaxel (60 mg/m2 for patients residing in East-Asian territories) given intravenously on Day 1 of each 21-day cycle.
  or 35 mg/m2 docetaxel given intravenously on a weekly basis as part of a continuous 21-day cycle; i.e. dosing will be on Days 1, 8, and 15 of each 21-day cycle.
  Treatment duration until radiographically confirmed disease progression.
Period: Overall Study
Arm/Group | Rociletinib 500 mg BID | Rociletinib 625 mg BID | Chemotherapy
Started | 53 | 22 | 74
Crossed Over to Rociletinib 500 mg BID | 0 | 0 | 36
Crossed Over to Rociletinib 625 mg BID | 0 | 0 | 3
Completed | 0 (Patients who are off study for any reason.) | 0 (Patients who are off study for any reason.) | 0 (Patients who are off study for any reason.)
Not Completed | 53 | 22 | 74
Not completed — Progressive Disease | 42 | 14 | 49
Not completed — Adverse Event | 3 | 4 | 6
Not completed — Death | 3 | 3 | 3
Not completed — Withdrawal by Subject | 1 | 1 | 6
Not completed — Physician Decision | 2 | 0 | 5
Not completed — Study Terminated by Sponsor | 2 | 0 | 0
Not completed — Missing | 0 | 0 | 1
Not completed — Miscellaneous | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rociletinib 500 mg BID | Rociletinib 625 mg BID | Chemotherapy | Total
Number analyzed (Participants) | 53 | 22 | 74 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (11.66) | 63.4 (12.30) | 61.4 (9.84) | 61.8 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 13 | 39 | 87
  Male | 18 | 9 | 35 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 3 | 7
  Not Hispanic or Latino | 46 | 22 | 68 | 136
  Unknown or Not Reported | 3 | 0 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 23 | 6 | 30 | 59
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 2 | 0 | 3 | 5
  White | 24 | 15 | 38 | 77
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 4 | 0 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 24 | 15 | 38 | 77
  Asian | 23 | 6 | 30 | 59
  Non-White, Non-Asian | 6 | 1 | 6 | 13
Number of Previous Therapies [Median (Full Range); unit: Therapies] | 3.0 [1.0 to 8.0] | 3.0 [2.0 to 6.0] | 3.0 [0.0 to 13.0] | 3.0 [0.0 to 13.0]
Time Since Diagnosis of NSCLC [Mean (Standard Deviation); unit: Months] — Population: Information missing for one patient in the Chemotherapy treatment group.
  Months
    number analyzed (Participants) | 53 | 22 | 73 | 148
    (all) | 42.6 (35.54) | 37.5 (16.92) | 39.0 (25.10) | 40.1 (28.29)
History of CNS Metastases [Count of Participants; unit: Participants] | 23 | 9 | 31 | 63

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) According to RECIST Version 1.1 as Determined by Investigator Review (invPFS)
Description: PFS was calculated as 1+ the number of days from the date of randomization to documented radiographic progression as determined by the investigator, or death due to any cause, whichever occurs first. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.The appearance of one or more new lesions is also considered progression.
Time Frame: Cycle 1 Day 1 to End of Treatment, up to approximately 35 months. This Time Frame includes the cross-over period, however, participants who crossed over to rociletinib were not analyzed for PFS.
Population: Intent-to-treat: All patients randomized. 1 patient in the Chemotherapy treatment group was not included in the analysis, due to discontinuation of study shortly after randomization and prior to first dose of study drug.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Rociletinib 500 mg BID | Rociletinib 625 mg BID | Chemotherapy
Number analyzed (Participants) | 53 | 22 | 73
Days | 125.0 [79.0 to 165.0] | 166.0 [56.0 to 246.0] | 77.0 [42.0 to 88.0]

2. Secondary Outcome: Percentage of Participants With Confirmed Response
Description: Percentage of patients with a best overall confirmed response of partial response (PR) or complete response (CR) recorded from the start of the treatment until disease progression or recurrence. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions, defined by and assessed as: Complete Response (CR), is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial Response (PR),at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameter. Overall Response (OR),is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The patient's best response assignment was dependent on the achievement of both measurement and confirmation criteria.
Time Frame: Cycle 1 Day 1 to End of Treatment, up to approximately 35 months. This Time Frame includes the cross-over period, however, participants who crossed over to rociletinib were not analyzed for best overall confirmed response.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rociletinib 500 mg BID | Rociletinib 625 mg BID | Chemotherapy
Number analyzed (Participants) | 53 | 22 | 73
percentage of participants | 17.0 [8.1 to 29.8] | 18.2 [5.2 to 40.3] | 8.2 [3.1 to 17.0]

3. Secondary Outcome: Duration of Response (DOR) According to RECIST Version 1.1 as Determined by Investigator Assessment
Description: DOR in patients with confirmed response per investigator. The DOR for complete response (CR) and partial response (PR) was measured from date that any of these best responses is first recorded until first date that progressive disease (PD) is objectively documented. For patients who continue treatment post-progression, the first date of progression was used for the analysis. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions, defined by and assessed as: CR is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10mm. PR is at least a 30% decrease in sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameter. Overall Response is the best response from start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Time Frame: Cycle 1 Day 1 to End of Treatment, up to approximately 35 months
Population: The DOR was measured only in those patients with a confirmed Complete Response (CR) or Partial Response (PR). The overall number of participants analyzed in the "Chemotherapy" arm includes only participants treated with chemotherapy and not patients who crossed over into the rociletinib treatment groups.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Rociletinib 500 mg BID | Rociletinib 625 mg BID | Chemotherapy
Number analyzed (Participants) | 9 | 4 | 6
Days | 335.0 [77.0 to 418.0] | 275.0 [167.0 to 375.0] | 206.0 [136.0 to NA] — Upper confidence limit is not available because it could be calculated.

4. Secondary Outcome: Overall Survival (OS)
Description: OS was calculated as 1+ the number of days from randomization to death due to any cause. Patients without a documented date of death were censored on the date the patient was last known to be alive.
Time Frame: Cycle 1 Day 1 to date of death, assessed up to 3 years
Population: Intent-to-treat: All patients randomized.1 patient in the Roci 500 and 2 patients in the Chemo treatment group were not included in the analysis because their OS data was not collected. 1 additional patient in the Chemo group was not included due to discontinuation from study shortly after randomization and prior to first dose of study drug.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Rociletinib 500 mg BID | Rociletinib 625 mg BID | Chemotherapy
Number analyzed (Participants) | 52 | 22 | 71
Days | 665 [232 to NA] — The upper Confidence Limit is not available because it could not be calculated. | 541 [173 to NA] — The upper Confidence Limit is not available because it could not be calculated. | 348 [231 to 522]

5. Secondary Outcome: Plasma PK for Patients Treated With Rociletinib Based on Sparse Sampling
Description: Blood samples were drawn for PK analysis at 21 ± 3 day intervals for the first 6 months (Day 1 of Cycles 2 to 7 inclusive). The sample could be taken predose or postdose. Plasma concentrations are presented for Rociletinib and 3 metabolites (M460, M502, M544).
Time Frame: Cycles 2 Day 1 to Cycle 7 Day 1, or approximately 6 months
Population: A small subset of patients treated with rociletinib (ie, patients randomized to receive rociletinib or who crossed over to receive rociletinib following treatment with single agent cytotoxic chemotherapy). Note: 2 patients in the 625mg treatment group had M502 values at upper limit of quantification (ULOQ) which were set as missing values.
Measure: Median (Full Range); unit: Plasma concentration (ng/mL)
Units Other Than Participants: Plasma samples
Arm/Group | Rociletinib 500 mg BID | Rociletinib 625 mg BID
Number analyzed (Participants) | 1 | 10
Number analyzed (Plasma samples) | 1 | 33
Plasma concentration (ng/mL)
  Rociletinib | 80.4 [80.4 to 80.4] | 207.0 [10.0 to 988.0]
  M460 | 20.0 [20.0 to 20.0] | 555.0 [144.0 to 1200.0]
  M502: number analyzed (Plasma samples) | 1 | 31
  M502 | 573.0 [573.0 to 573.0] | 3260.0 [98.4 to 4880.0]
  M544 | 765.0 [765.0 to 765.0] | 525.0 [20.0 to 3640.0]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the date of first dose of study drug and within 28 days after last dose of study drug, an average of 6 months. In addition, study procedure-related AEs that occur after signing of the informed consent form and before first dose of study drug were expected to be reported. Any Serious Adverse Events or Adverse Events of Special Interest were followed until resolution or stabilization, or until patient is lost to follow-up.
Description: If a subject experiences the same preferred term (system organ class) multiple times, then the subject will be counted only once for that preferred term (system organ class). Treatment Arm/Groups for subjects who crossed over to Rociletinib from Chemotherapy are included. 1 patient in the Chemotherapy treatment group was not included in the analysis, due to discontinuation of study shortly after randomization and prior to first dose of study drug.
Groups:
- Rociletinib 500 mg BID: Starting dose of 500 mg. Taken orally twice daily (continuous 21 day treatment cycle). Treatment duration until radiographically confirmed disease progression.
- Rociletinib 625 mg BID: Starting dose of 625 mg. Taken orally twice daily (continuous 21 day treatment cycle). Treatment duration until radiographically confirmed disease progression.
- Crossover From Chemotherapy to Rociletinib 500 mg BID: Patients initially randomized to comparator chemotherapy had the option to cross over to rociletinib following disease progression per RECIST Version 1.1. Rociletinib starting dose of 500 mg taken orally twice daily (continuous 21 day treatment cycle). Treatment duration until radiographically confirmed disease progression.
- Crossover From Chemotherapy to Rociletinib 625 mg BID: Patients initially randomized to comparator chemotherapy had the option to cross over to rociletinib following disease progression per RECIST Version 1.1. Rociletinib starting dose of 625 mg taken orally twice daily (continuous 21 day treatment cycle). Treatment duration until radiographically confirmed disease progression
Arm/Group | Rociletinib 500 mg BID | Rociletinib 625 mg BID | Chemotherapy | Crossover From Chemotherapy to Rociletinib 500 mg BID | Crossover From Chemotherapy to Rociletinib 625 mg BID
All-Cause Mortality (participants affected / at risk) | 10/53 | 3/22 | 3/73 | 6/36 | 0/3
Serious Adverse Events (participants affected / at risk) | 23/53 | 7/22 | 23/73 | 18/36 | 1/3
Other Adverse Events (participants affected / at risk) | 53/53 | 21/22 | 71/73 | 35/36 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rociletinib 500 mg BID (N=53) | Rociletinib 625 mg BID (N=22) | Chemotherapy (N=73) | Crossover From Chemotherapy to Rociletinib 500 mg BID (N=36) | Crossover From Chemotherapy to Rociletinib 625 mg BID (N=3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardio-pulmonary arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 3 | 0
Generalised oedema (General disorders) | 1 | 0 | 0 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 1 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Intervertabral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1 | 2 | 2 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0
Complex partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Nodal arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 2 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rociletinib 500 mg BID (N=53) | Rociletinib 625 mg BID (N=22) | Chemotherapy (N=73) | Crossover From Chemotherapy to Rociletinib 500 mg BID (N=36) | Crossover From Chemotherapy to Rociletinib 625 mg BID (N=3)
Anaemia (Blood and lymphatic system disorders) | 7 | 2 | 18 | 5 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 5 | 4 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 9 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 5 | 2 | 0
Cataract (Eye disorders) | 5 | 3 | 1 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 0 | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 6 | 2 | 10 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 33 | 15 | 12 | 13 | 1
Dry mouth (Gastrointestinal disorders) | 3 | 1 | 2 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 5 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 2 | 2 | 2 | 0
Nausea (Gastrointestinal disorders) | 19 | 9 | 20 | 7 | 1
Stomatitis (General disorders) | 3 | 1 | 4 | 0 | 0
Vomiting (Gastrointestinal disorders) | 10 | 8 | 6 | 6 | 2
Asthenia (General disorders) | 10 | 1 | 10 | 3 | 0
Chest discomfort (General disorders) | 3 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 2 | 2 | 0 | 0
Fatigue (General disorders) | 16 | 12 | 18 | 4 | 1
Non-cardiac chest pain (General disorders) | 3 | 0 | 5 | 3 | 0
Oedema peripheral (General disorders) | 5 | 1 | 6 | 1 | 0
Pyrexia (General disorders) | 5 | 2 | 7 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 2 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 3 | 0 | 0
Urinary tract infection (Infections and infestations) | 4 | 1 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 2 | 4 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 1 | 5 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 0 | 3 | 1 | 0
Blood bilirubin increased (Investigations) | 4 | 4 | 1 | 2 | 0
Blood creatinine increased (Investigations) | 4 | 1 | 3 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 10 | 10 | 0 | 7 | 1
Lymphocyte count decreased (Investigations) | 2 | 1 | 4 | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 0 | 10 | 0 | 0
Platelet count decreased (Investigations) | 3 | 1 | 4 | 0 | 0
Weight decreased (Investigations) | 10 | 4 | 4 | 1 | 1
White blood cell count decreased (Investigations) | 2 | 3 | 9 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 19 | 9 | 10 | 8 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 30 | 14 | 6 | 12 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 6 | 3 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 2 | 4 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 3 | 2 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 0 | 6 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 3 | 10 | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 3 | 0 | 3 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 6 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 2 | 3 | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 3 | 2 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 4 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 1 | 2 | 2 | 1
Dizziness (Nervous system disorders) | 4 | 3 | 2 | 2 | 0
Headache (Nervous system disorders) | 6 | 5 | 5 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 4 | 0 | 0
Insomnia (Psychiatric disorders) | 8 | 1 | 10 | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 4 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 6 | 14 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 10 | 6 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 0 | 8 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 0 | 4 | 0 | 0
Hypertension (Vascular disorders) | 6 | 0 | 2 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 3 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0

LIMITATIONS AND CAVEATS:
Due to early study termination, only 149 of 600 planned patients were randomized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All parties agree to submit all manuscripts or abstracts to all other parties 30 days prior to submission. This will enable all parties to protect proprietary information and to provide comments based on information that may not yet be available to other parties. The sponsor may request a delay in publication if there are important intellectual property concerns relating to publication, but does not have the right to suppress publication of the study results indefinitely.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT02322281/Prot_SAP_000.pdf